CLINICAL TRIAL: NCT00123305
Title: A Multicentre, Double-Blind, Placebo-Controlled, Ascending-dose, Clinical Trial of Intravenous Microplasmin Administration in Patients With Acute Ischemic Stroke
Brief Title: Intravenous Administration of Microplasmin for Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-M-004
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Stroke, Acute
Keywords: Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Microplasmin
- 2 (Experimental)
  Interventions: Drug: Microplasmin
- 3 (Experimental)
  Interventions: Drug: Microplasmin
- 4 (Placebo Comparator)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — 1mg/kg bolus of microplasmin solution followed by 1,2 or 3mg/kg infusion of mircroplasmin solution.
  Arms: 1; 2; 3
Drug: Microplasmin — 1mg/kg bolus of placebo solution followed by 1,2 or 3mg/kg infusion of placebo solution
  Arms: 4

SUMMARY:
The primary purpose of this study is to evaluate the safety and preliminary efficacy of microplasmin when administered intravenously to patients who have suffered an acute stroke within 12 hours before randomization.

DETAILED DESCRIPTION:
While the primary objective of the trial is safety evaluation, efficacy assessments will also be obtained, including MRI/MRA (including DWI, PWI and T2 imaging) and plasma surrogate biomarkers. Clinical outcome will also be assessed at 7days, 30 days and 90 days post-treatment. At each of these visits, mortality and neurological assessments (NIHSS, Barthel index, mRankin scale) will be performed. In addition, vital status will be assessed vial a telephone contact at 60 days post-treatment.

The trial will investigate three dose regimens of microplasmin, all of which are within the range of doses previously evaluated in a Phase I trial in healthy volunteers; the planned sample size for the trial is approximately 40 patients.

The study will consist of 3 phases - the Baseline, In-hospital Phase and Follow up Phase. Baseline is from study entry through randomisation; the In-hospital phase is from treatment with study drug through hospital discharge or day 7, whichever occurs first. The follow up phase consists of visits to the hospital 30 days (+ 3 days) from the day of study drug administration. Hospital discharge is defined as the end of the discharge from the acute hospital setting. Discharge may be to home, to a rehabilitation setting or to a non-acute hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke with onset within 12 hours before randomization with baseline NIHSS > 6 and < 22

Exclusion Criteria:

General Exclusion Criteria

* Participation in another study with an investigational drug or device within the previous 30 days, prior participation in the present study, or planned participation in another trial within the time frame of the current trial
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan or MRI is negative for hemorrhage
* Women known to be pregnant, lactating, or having a positive or indeterminate pregnancy test

Stroke Related Exclusion Criteria

* Neurological deficit that has led to stupor or coma (National Institutes of Health Stroke Scale [NIHSS] Level Of Consciousness Item 1a score >or=2)
* High clinical suspicion of septic embolus
* Thrombosis involving cerebral veins
* Rapidly improving neurological signs at any time before initiation of study drug administration

Imaging Related Exclusion Criteria

* Hemorrhagic transformation or intracerebral hemorrhage observed on baseline CT of the brain or gradient recalled echo (GRE) magnetic resonance imaging
* CT or MRI evidence of nonvascular cause for the neurological symptoms
* Large hypodensity on CT involving > 1/3 of the middle cerebral artery (MCA) territory
* Baseline DWI volume > 1/3 of the MCA territory
* Signs of mass effect causing shift of midline structures on CT or MRI
* Unable to undergo MRI (i.e., ferrous implants, cardiac pacemakers, agitation, claustrophobia or known sensitivity to MRI contrast agents)

Safety Related Exclusion Criteria

* Congenital or acquired coagulopathy causing either of the following

  1. activated partial thromboplastin time prolongation greater than 2 seconds above the upper limit of normal (ULN) for local laboratory
  2. International normalized ratio (INR) of 1.4 or more.
* Uncontrolled hypertension defined as a systolic blood pressure > 180 mm Hg or a diastolic blood pressure > 100 mm Hg on 3 separate occasions at least 10 minutes apart or requiring continuous intravenous (IV) therapy.
* History of stroke within the previous 3 months
* Seizures at any time between stroke onset to planned initiation of study drug
* History of intracranial hemorrhage
* History of surgery, lumbar puncture, biopsy or trauma to internal organs within the previous 30 days.
* Major trauma at the time of stroke
* Head trauma within the previous 90 days.
* Known bleeding diathesis.
* Baseline platelet count < 100 X 10^9/L.
* Blood glucose > 400mg/dl or <50 mg/dl if administration of glucose does not rapidly reverse neurological deficit

Exclusion Criteria That May Potentially Interfere with Outcome Assessment

* Life expectancy <3 months
* Other serious illness that in the opinion of the investigator may confound clinical assessment (e.g. hepatic, cardiac, or renal failure, advanced cancer)

Exclusion Criteria Related to Concomitant Medication

* If treatment with tPA is indicated
* Treatment with rtPA or any other thrombolytic agent for the qualifying stroke
* Administration of intra-arterial or systemic thrombolytic therapy in previous 7 days
* Need for antiplatelet agent, unfractionated or heparin-related products, direct thrombin inhibitor, oral anticoagulant within 24 hours after treatment bolus.
* Treatment with low molecular weight heparin, direct thrombin inhibitor, or GPIIb/IIIa antagonists within 48 hours prior to randomisation
* Treatment with vitamin-K antagonists or heparin (or heparin-related compounds) which results in either an INR>1.4 or an aPTT>2 times control (ULN for the hospital laboratory)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Intracranial haemorrhage | 24 hours and Day-7
Change from Baseline in NIHSS | Day7 and Day-90

SECONDARY OUTCOMES:
Barthel Index and modified Rankin scale | Day-90
Markers of systemic lysis | Baseline, end of treatment, 6, 12, 24, 72 and 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Thijs, MD PhD, Principal Investigator — KU Leuven
Locations (16):
- Austria (4):
  - Universitatsklinik fur Neurologie, Graz
  - Landesnervenklinik Wagner-Jauregg, Linz
  - AKH Linz Neurolog Abt, Linz
  - Allgemeines Offentliches Krankenhaus der, Linz
- Belgium (2):
  - Cliniques Universitaires St Luc, Brussels
  - Gasthuisburg Hospital, Leuven
- Germany (10):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - Klinikum der J.W Goethe Univeristy, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Georg August Universitat Gottingen, Göttingen
  - Universitatskrankenhaus Hamburg-Eppendorf, Hamburg
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Minden, Chefarzt der Neurologischen Klinik, Minden
  - Klinikum rechts der Isar der TU München, München
  - HSK Dr. Horst Schmidt Hospital, Wiesbaden